CLINICAL TRIAL: NCT04879979
Title: Cognitive Impairment in GIST Patients on Tyrosine Kinase Inhibitor Therapy: Cognitive Behavioral Therapy to Improve Cognitive Symptoms
Brief Title: GIST and Memory and Attention Adaptation Training
Acronym: GIST-MAAT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Robert J Ferguson, PhD, Assistant Professor of Medicine, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HCC 20-117
Record Dates: First submitted 2021-04-28; First posted 2021-05-10 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: GIST, Malignant; CBT
Keywords: GIST; MAAT; CBT
MeSH Terms: conditions — Gastrointestinal Stromal Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Memory and Attention Adaptation Training (MAAT) (Experimental): A cognitive-behavioral therapy (CBT) designed for the treatment of Cancer-Related Cognitive Impairment (CRCI)
  Interventions: Behavioral: MAAT

INTERVENTIONS:
Behavioral: MAAT — MAAT consists of 8 weekly visits of 45 minutes duration and can be delivered effectively through videoconference technology (Vidyo). Participants will be asked to download the Vidyo App on their mobile phone or tablet. Vidyo is a HIPPA compliant, encrypted software with adequate bandwidth for highest quality videoconferencing intended for telehealth. It is the primary software for UPMC Telemedicine. Survivors are provided a workbook to reinforce learning, mastery and application of skills in daily life covered in each MAAT visit. The workbook provides reading structured within each of the 8 visits with guides for application of strategies as homework

SUMMARY:
Cognitive-behavioral therapy (CBT) has been found to be efficacious in the treatment of cancer-related cognitive impairment (CRCI). Memory and Attention Adaptation Training (MAAT) has been evaluated in previous clinical trials with samples of breast cancer survivors and found effective at reducing cancer-related cognitive impairment. MAAT has been demonstrated to be efficacious when it is delivered via videoconference.The use of telehealth delivery enhances access to cancer survivorship care and reduces time and travel burden among cancer survivors, especially those who live in rural and/or underserved areas where cancer survivor services are less available.

People with a diagnosis of gastrointestinal stromal tumors also experience self-reported cancer-related cognitive impairment. In order to determine if MAAT can sufficiently treat CRCI among people with gastrointestinal stromal tumors (GIST), we propose a trial of MAAT to determine its initial level of effectiveness in improving both self-reported cognitive impairments and objective neuropsychological test performance in GIST patients.

DETAILED DESCRIPTION:
This study is a single-group, repeated measures (pre-post-intervention) design. This low-cost, simple design is intended to gather pilot data to gain an understanding of preliminary MAAT efficacy in the population of people with GIST who have cognitive complaints. The objective of the study is to estimate the magnitude of clinical effect of MAAT (delivered via videoconference, telehealth technology) on perceived cognitive impairment and neuropsychological test performance among GIST patients with cognitive complaints. The primary objectives consist of the telephone-based assessment of neuropsychological status (TBANS) and self-reported cognitive symptoms as assessed by the FACT-Cog perceived cognitive impairments (PCI) scale and impact on quality of life scale (IQOL). Within-group effect size will be calculated to determine clinical effect of MAAT on group outcomes on neuropsychological and self-reported outcome measures (PCI, IQOL). The reliable change index (RCI) will be calculated to determine minimal clinically important differences in pre-to-post change in individual cases on FACT-Cog (PCI; IQOL) outcomes. The proportion of cases who exceed reliable change ("reliable" difference in pre-to-post-intervention FACT-Cog scores) will be quantified. The secondary objective is to estimate the magnitude of effect of MAAT on depressive symptoms, anxiety and fatigue among GIST patients with cognitive complaints. This will be done using a self-reported questionnaire (total scores/T-scores); a within-group effect size calculated to determine clinical effect of MAAT on group outcomes on self-reported outcome measures (PROMIS Depression 8a; PROMIS Anxiety 8a, PROMIS® Pain 3a, PROMIS® Fatigue 8a) and a within group effect size to determine clinical effect on group outcomes and published minimal clinically important differences in pre-to-post change individual cases. Screening will begin with individual patients diagnosed with GIST and who have either been directed by medical oncologists or those who respond to advertisements on clinic video monitors in waiting rooms, or who have responded to Pitt+Me recruitment methods. All participants in this study will be able to participate from home through the telephone (pre-post-MAAT, or intervention, neurocognitive assessments) and mobile device telehealth videoconference visits for 8 MAAT visits (intervention). Eligible and consented participants will have their first telephone-based neurocognitive assessment (TBANS) scheduled shortly after consent. At that point, a trained psychometrist (our research coordinator) will schedule the 30-minute telephone based and standardized neurocognitive assessment. Participants will also complete self-report measures online (REDCap) with data stored on secured University of Pittsburgh servers.Participants will then be enrolled in MAAT for 8 weekly visits of 45minutes each (described below). MAAT will be videoconference delivered by doctoral-level clinical psychology graduate student trainees who will be completing clinical externship with the Center for Counseling and Cancer Support at Hillman Cancer Center, Shadyside Medical Building. Dr. Ferguson will train and supervise each trainee delivering MAAT to assure highest quality control and treatment fidelity. After completion of 8 MAAT visits, participants will complete post-intervention measures consisting of the same measures they performed during the pre-intervention excluding demographic, clinical characteristics, and Charlson Comorbidity Index to evaluate participant change (efficacy) due to MAAT intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 and above;
2. Diagnosis of Gastrointestinal stromal tumor (GIST);
3. At least 1 year post-initiation of TKI therapy;
4. Report cognitive problems of memory and concentration attributed to GIST and/or treatment with a score of 10 or below on the FACT-Cog Impact on Quality of Life Scale;
5. Able to speak and read English;
6. Able to provide IRB-approved written informed consent; and
7. Willingness to use videoconferencing and complete phone-based neurocognitive assessments

Exclusion Criteria:

1. Previous treatment with a tyrosine kinase inhibitor medication for a non-GIST diagnosis
2. Previous CNS radiation, intrathecal therapy, or CNS-involved surgery;
3. Previous cancer history with the exception of non-melanoma skin cancer;
4. Previous exposure to chemotherapy with another cancer or due to other medical condition (e.g., methotrexate exposure for treatment of rheumatoid arthritis);
5. Scoring 3 or below on the 6-item cognitive screen designed to detect severe memory disorders;1
6. Significant neurodevelopmental, neurobehavioral, or medical risk factors likely to affect cognitive functioning (e.g., history of neurological disorder, stroke, traumatic brain injury greater than mild severity, such as loss of consciousness >30 minutes, medical disorder that is unstable or likely to affect cognition such as metabolic disorder, heart attack, uncontrolled diabetes or endocrine dysfunction);
7. Current severe DSM-5 mental disorder criteria, including but not limited to neurodevelopmental, substance abuse, mood, anxiety, or psychotic disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-01-12 (Actual); Primary Completion 2022-05-04 (Actual); Study Completion 2022-05-04 (Actual)

PRIMARY OUTCOMES:
California Verbal Learning Test-3 (CVLT-3) | After 8 weekly MAAT visits (or up to 12 weeks if weekly visits are rescheduled)
  The California Verbal Learning Test is a neuropsychological assessment of episodic verbal and working memory. Participants listen to series of words and are then asked to recall the terms and the category to which they belong. This assessment attempts to measure how much a subject learned and also reveal strategies employed and the types of errors made. CVLT-3 measures both recall and recognition of two lists of words (List A and List B). Higher CVLT-3 scores (number of words recalled) are associated with better memory and processing function, therefore better outcome. Scores range from 0-16 for each word list where the higher the score the better the outcome.
Controlled Oral World Association Test (COWAT) | After 8 weekly MAAT visits (or up to 12 weeks if weekly visits are rescheduled)
  The Controlled Oral Word Association Test (COWAT), is a neuropsychological measure of verbal fluency. The COWAT consists of three word conditions. Participants are asked to produce as many words as they can that begin with the F, A, or S within a 1 minute time period. The total number of words that the individual is able to produce provides a score.
Symbol Digit Modalities Test (SDMT) | After 8 weekly MAAT visits (or up to 12 weeks if weekly visits are rescheduled)
  The Symbol Digit Modalities Test (SDMT) is a neurocognitive screening instrument used to assess neurological dysfunction. Participants are required to use a coded key to match nine abstract symbols paired with numerical digits. Ten (10) practice items before commencing the test. The final score is the correct number of substitutions in 90 seconds, and scores range between 0 and 110. Higher scores indicate better neurocognitive functioning.

SECONDARY OUTCOMES:
FACT-Cog PCI | After 8 weekly MAAT visits (or up to 12 weeks if weekly visits are rescheduled)
  The FACT-Cog is a 37-item self-report measure that uses 5- point (0-4) Likert-type ratings that produce four scales: 1) Impact on quality of life; 2) Perceived cognitive impairments; 3) Comments from others; and 3) Perceived cognitive abilities. Higher scores indicate better function and quality of life on each scale. While each scale is scored and interpreted separately, they comprise the total Fact-cog assessment.
PROMIS Item Bank -Emotional Distress - Short Form 8a | After 8 weekly MAAT visits (or up to 12 weeks if weekly visits are rescheduled)
  This measure assesses self-reported negative mood, views of self, and social cognition, as well as decreased positive affect and engagement. It has 8 items on a 5-pt Likert Scale (1-5). Scores range from 8-40, where higher scores indicate more emotional distress.
PROMIS Item Bank: Anxiety- Short Form 8a. | After 8 weekly MAAT visits (or up to 12 weeks if weekly visits are rescheduled)
  Measures self-reported fear (fearfulness, panic), anxious misery (worry, dread), and hyperarousal (tension, nervousness, restlessness). It contains 8 items on a 5-pt Likert Scale (1-5). Scores range from 8-40, where higher scores indicate higher levels of anxiety.
PROMIS Short Form: Fatigue 8a. | After 8 weekly MAAT visits (or up to 12 weeks if weekly visits are rescheduled)
  Assesses subjective symptoms of fatigue from mild subjective feelings of tiredness to a sustained sense of exhaustion that interferes with function. It contains 8 items on a 5-pt Likert scale (1-5). Scores range from 8-40 where higher scores indicate higher levels of fatigue.
PROMIS Short Form: Pain 3a. | After 8 weekly MAAT visits (or up to 12 weeks if weekly visits are rescheduled)
  Assesses worst, average and current pain intensity. It contains 3 items on a 5 point Likert scale (1-5). Scores range from 3-15, where higher scores indicate higher levels of pain.

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Ferguson, PhD, Principal Investigator — University of Pittsburgh School of Medicine, UPMC Hillman Cancer Center; Anette U Duensing, MD, Principal Investigator — University of Pittsburgh School of Medicine, UPMC Hillman Cancer Center
Locations (1):
- UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No